CLINICAL TRIAL: NCT02863809
Title: A Phase I/II Prospective, Randomized, Multicenter, Double-Masked, Vehicle-Controlled Clinical Trial to Evaluate the Safety and Efficacy of Corneal Collagen Cross-Linking of Keratoprosthesis Carrier Tissue in High-Risk Keratoprosthesis Implantation
Brief Title: Vision Restoration With a Collagen Crosslinked Boston Keratoprosthesis Unit
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joseph B. Ciolino, MD (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Joseph B. Ciolino, MD, Professor of Opthalmology, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 798474
Record Dates: First submitted 2016-06-01; First posted 2016-08-11 (Estimated); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Keratolysis
Keywords: Keratolysis; Corneal Melting; Boston KPro; Keratoprosthesis
MeSH Terms: interventions — Riboflavin; Dextrans; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Active Treatment Arm (Experimental): De-epithelialized corneas cross-linked with riboflavin 0.1% and dextran 20% solution AND ultraviolet A light (UVA Light Source).
  Interventions: Drug: Riboflavin; Drug: Dextran; Device: UVA Light Source
- Control Treatment Arm (Active Comparator): De-epithelialized corneas will be exposed to only riboflavin 0.1% with dextran 20% solution (NO ultraviolet A light).
  Interventions: Drug: Riboflavin; Drug: Dextran

INTERVENTIONS:
Drug: Riboflavin — Riboflavin, a water soluble vitamin, is an essential nutrient and a natural component of many foods.
  Other Names: Vitamin B2
Drug: Dextran — Dextran is used to increase the viscosity of the solution.
  Other Names: Dextran 70 6% in 0.9%; Sodium Chloride Dextran 70 6% in 5% Dextrose; Gentran 70, Hyskon
Device: UVA Light Source — Avedro's KXL® System is a UVA irradiation system that uses a light emitting diode (LED) to deliver a dose of UVA light to a targeted treatment area for illuminating the cornea during corneal collagen cross-linking.
  Other Names: KXL® System
  Arms: Active Treatment Arm

SUMMARY:
This is a phase I/II prospective, randomized, multi-center, double-masked, vehicle-controlled clinical trial evaluating the safety and efficacy of corneal collagen cross-linking the keratoprosthesis carrier tissue in subjects who are candidates for high-risk keratoprosthesis implantation but because of a history of corneal melts or autoimmune diseases are not candidate for a traditional corneal transplant.

DETAILED DESCRIPTION:
The study is a multi-center, parallel, randomized, double-blinded study with subsequent follow-up period of two years. Eight-four subjects across twelve sites will be randomized 1:1 to receive either a corneal tissue that have been cross-linked or not cross-linked (No UVA light source). Cross-linking is a term that refers to the linking of polymers (long chain) molecules by chemical bonds. It is believed that cross-linking the cornea will make the cornea stronger and more resistant to degradation.

CorneaGen (formerly Keralink International) (Baltimore site) will supply the donor tissue and Avedro Inc (Waltham MA) will supply the riboflavin and the UV light source. Staff at CorneaGenwill administer the riboflavin with dextran solution and perform the cross-linking procedure according to one of randomization groups before shipping the masked donor cornea to study sites for Boston Keratoprosthesis (B-KPro) implantation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Willing and able to comply with study assessments for the full duration of the study
* Age ≥ 18 years
* Candidate for a Boston Keratoprosthesis / Cornea transplant
* In generally good stable overall health
* Patients with an eye at risk for a cornea sterile ulcer which includes:

  * Autoimmune diseases (mucus membrane pemphigoid, Stevens-Johnson syndrome, systemic lupus erythematosis, rheumatoid arthritis, or other autoimmune diseases); OR
  * History of previous sterile cornea ulceration requiring a cornea transplant

Exclusion Criteria:

* Age < 18 years
* Inability to provide written informed consent and comply with study assessments for the full duration of the study
* No or minimal tear production with evidence of keratinization of the bulbar conjunctiva
* Corneal or ocular surface infection within 30 days prior to study entry
* Ocular or periocular malignancy
* Inability to wear a contact lens due to lid abnormalities or shortened fornix
* Signs of current infection, including fever and current treatment with antibiotics
* Pregnancy (positive pregnancy test) or lactating
* Participation in another simultaneous interventional medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B. Ciolino, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (13):
- United States (13):
  - The Jules Stein Eye Institute, Los Angeles, California
  - UC Davis Health System Eye Center, Sacramento, California
  - Shiley Eye Institute, University of California, San Diego, San Diego, California
  - Bascom Palmer eye Institute, Miami, Florida
  - Illinois Eye and Ear Infirmary, Chicago, Illinois
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Wilmer Eye Institute, Baltimore, Maryland
  - W.K. Kellogg Eye Center, Ann Arbor, Michigan
  - Tauber Eye Center, Kansas City, Missouri
  - David and Ilene Flaum Eye Institute, University of Rochester, New York, New York
  - University Hospitals Eye Institute, Cleveland, Ohio
  - Wills Eye, Bala-Cynwyd, Pennsylvania
  - Wilford Hall Ambulatory Surgical Center (WHASC), Lackland Air Force Base, Texas

IPD SHARING:
Plan to Share IPD: No
The data within StudyTrax will be extracted at the completion of the study. This data will be held in a secure network file at MEEI for at least two years following a marketing application submission to the FDA or longer, if required by the MEEI IRB.

REFERENCES:
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 76 subjects enrolled - signed consent form
  * 5 screen fails (did not meet eligibility criteria);
  * 1 withdrawal (signed consent form but declined to participate before randomization occurred)
  * 2 other (signed consent forms but were not able to receive surgery due to COVID-19 restrictions)
Period: Overall Study
Arm/Group | Active Treatment Arm | Control Treatment Arm
Started (Subjects randomized in the study groups) | 34 | 34
Screen Fail (Post Randomization) (Subject that did not meet eligibility criteria after the study randomization had occured.) | 1 | 0
Completed | 24 | 24
Not Completed | 10 | 10
Not completed — Adverse Event | 8 | 8
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants receiving cross-linked (CXL) versus non-cross-linked (non-CXL) donor corneas (One subject who was randomized in the active arm (CXL corneal carrier) was excluded from efficacy analysis due to not meeting the inclusion criteria)
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment Arm | Control Treatment Arm | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (15.3) | 62.8 (16.9) | 62.3 (15.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 20 | 23 | 43
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Previous sterile keratolysis [Count of Participants; unit: Participants] | 28 | 28 | 56
Autoimmune disease [Count of Participants; unit: Participants]
  Steven Johnson Syndrome | 3 | 4 | 7
  Rheumatoid Arthritis | 1 | 3 | 4
  Graft Versus Host Disease | 1 | 1 | 2
  Mucus Membrane Pemphigoid | 1 | 0 | 1
  Vogt-Koyangi-Harada Syndrome | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time From Surgery to Device Loss or Replacement
Description: If the device fails after surgery the time and reason behind the failure will be recorded. The number of device losses in the control group will be compared to the number of device losses in investigational group.
Time Frame: 2 years
Measure: Median (Inter-Quartile Range); unit: median weeks from surgery to removal
Arm/Group | Active Treatment Arm | Control Treatment Arm
Number analyzed (Participants) | 33 | 34
median weeks from surgery to removal | 95 [60 to 117] | 34 [11 to 66]

2. Secondary Outcome: Number of Participants With Kpro Retention at 12 Months
Description: The number of participants that retained kpro devices at the end of twelve months will be studied and differences in retention rate between investigational and control groups will be reported
Time Frame: Twelve months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Arm | Control Treatment Arm
Number analyzed (Participants) | 33 | 34
Participants | 29 | 27

3. Secondary Outcome: Number of Cumulative Delayed Epithelial Healing Events at Day 30
Description: The number of incidences of delayed epithelial healing at day 30 will be recorded. If there is delayed epithelial healing at day 30 it will be determined if those incidences occurred more often in the control group versus the investigational group.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Arm | Control Treatment Arm
Number analyzed (Participants) | 33 | 34
Participants | 10 | 10

4. Secondary Outcome: Median Time From Surgery to Retroprosthetic Membrane Treatment in Days (Laser or Surgical Interventions)
Description: If follow up surgery is needed to replace or treat the prosthetic the time and reason will be recorded and the number of incidences will be compared between the study treatment groups
Time Frame: 2 years
Measure: Median (Standard Deviation); unit: median time (days) from surgery to RPM
Arm/Group | Active Treatment Arm | Control Treatment Arm
Number analyzed (Participants) | 33 | 34
median time (days) from surgery to RPM | 300.3 (194.7) | 253.37 (158.11)

5. Secondary Outcome: Median Time From Surgery to Occurrence of Vitritis (Sterile or Infectious)
Description: The time (days) and number of incidences of vitritis will be recorded for the subject in which it occurred and the number of incidences will be compared between the study treatment groups.
Time Frame: 2 years
Measure: Median (Standard Deviation); unit: median time (days) surgery to vitritis
Arm/Group | Active Treatment Arm | Control Treatment Arm
Number analyzed (Participants) | 33 | 34
median time (days) surgery to vitritis | 188.6 (218.4) | 254.3 (239.6)

ADVERSE EVENTS:
Time Frame: Day 1, Week 1, Week 4, Week 16, Week 36, Week 52, Week 78, Week 104, Week 130, Week 156, Week 182
Description: Adverse Event - Any untoward or unfavorable medical occurrence in a human subject. Only adverse events that met a frequency threshold of 5% have been reported to CT.gov (occurred in greater than 5% of the study participants).
  Serious Adverse Event - For this study, a Serious Adverse Event is defined as any event temporally associated with the subject's participation in research that results in death; is life threatening; requires hospitalization;
Arm/Group | Active Treatment Arm | Control Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 6/34 | 10/34
Other Adverse Events (participants affected / at risk) | 17/34 | 16/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment Arm (N=34) | Control Treatment Arm (N=34)
Infection (Eye disorders) | 2 (2) | 1 (1) — 1. Possible infectious keratitis 2. Infection of glaucoma bleb (blebitis and endophthalmitis)
Corneal Melt (Eye disorders) | 2 (2) | 3 (3) — Corneal Melt
High Intraocular Pressure (Eye disorders) | 0 (0) | 1 (2) — High Intraocular Pressure
Choroidal Detachment (Eye disorders) | 1 (2) | 0 (0) — Choroidal Detachment
Endophthalmitis (Eye disorders) | 1 (1) | 0 (0) — Endophthalmitis (right eye)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1)
Complication of corneal transplant (Eye disorders) | 0 (0) | 1 (1) — Complication of corneal transplant (gap between front plate and donor)
Persistent Epithelial Defect (Eye disorders) | 0 (0) | 1 (1) — Persistent Epithelial Defect
Epiretinal membrane (Eye disorders) | 0 (0) | 1 (1) — Epiretinal membrane
Wound Dehiscence (Eye disorders) | 0 (0) | 1 (1) — Wound Dehiscence
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment Arm (N=34) | Control Treatment Arm (N=34)
Retroprosthetic Membrane (Eye disorders) | 4 (4) | 3 (4) — Retroprosthetic Membrane
Vitreous (Eye disorders) | 2 (4) | 5 (5) — Vitreous hemorrhage
Corneal Thinning (Eye disorders) | 1 (1) | 2 (2) — Corneal thinning
EPI Defect (Eye disorders) | 3 (3) | 3 (4) — Epi defect
High Intraocular Pressure (Eye disorders) | 2 (2) | 2 (2) — High Intraocular Pressure
Eye Pain (discomfort) (Eye disorders) | 2 (4) | 3 (3) — Eye Pain (discomfort)
Loose suture (Eye disorders) | 2 (4) | 1 (1) — Loose suture
Hemmorrge (Eye disorders) | 3 (3) | 0 (0) — Hemmorrge

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT02863809/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT02863809/SAP_002.pdf